CLINICAL TRIAL: NCT00482521
Title: A Phase I, Open-Label Study to Determine the Maximum Tolerated Dose (MTD) and to Evaluate the Safety Profile of CC-4047 in Subjects With Advanced Solid Tumors
Brief Title: CC-4047 in Treating Patients With Advanced Solid Tumors That Did Not Respond to Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE4Y06; P30CA043703 (NIH); CASE4Y06 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2007-06-04; First posted 2007-06-05 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2012-08

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CC-4047 (Experimental)
  Interventions: Drug: CC-4047

INTERVENTIONS:
Drug: CC-4047 — Oral CC-4047 once daily on days 1-21 followed by a 7-day recovery period. Cohorts of 3-6 patients receive escalating doses of CC-4047 until the maximum tolerated dose (MTD) is determined.

SUMMARY:
RATIONALE: CC-4047 may stop the growth of tumor cells by blocking blood flow to the tumor.

PURPOSE: This phase I trial is studying the side effects and best dose of CC-4047 in treating patients with advanced solid tumors that did not respond to treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of CC-4047 in patients with advanced refractory solid tumors.

Secondary

* Assess the safety of this drug in these patients.
* Assess the antitumor activity of this drug in these patients.
* Determine the effect of this drug on fetal hemoglobin levels in these patients.

OUTLINE: This is a open-label, uncontrolled, nonrandomized, dose-escalation, multicenter study.

* Treatment phase (course 1): Patients receive oral CC-4047 once daily on days 1-21 followed by a 7-day recovery period.

Cohorts of 3-6 patients receive escalating doses of CC-4047 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity (DLT).

Patients with no clinical evidence of progressive disease or DLT after course 1 continue study treatment during the extension phase. Patients who develop a DLT during course 1 may continue study treatment at the discretion of the investigator.

* Extension phase: Patients continue taking CC-4047 at their assigned cohort dose as in course 1. Patients who tolerate a treatment-phase dose higher than the MTD continue treatment at the MTD. Courses repeat every 28 days for up to 24 months in the absence of disease progression or unacceptable toxicity.

Patients undergo blood collection at baseline and periodically during study to evaluate fetal hemoglobin levels.

After completion of study treatment, patients are followed at 28 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced solid tumor
* Refractory disease

  * Patients must have been offered and refused OR received and failed prior treatment with all standard or approved therapies for the malignancy
* Measurable or evaluable disease as confirmed by radiographic or clinical evidence
* No curative therapy available

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 3 months
* ANC > 1,500/mm³
* Platelet count > 75,000/mm³
* Hemoglobin ≥ 9.0 g/dL
* Creatinine ≤ 2.0 mg/dL
* AST and ALT < 3 times upper limit of normal
* Not pregnant
* No nursing during and for ≥ 28 days after completion of study treatment
* Two negative pregnancy tests required
* Fertile women must use effective double-method contraception for ≥ 28 days before, during, and for ≥ 28 days after completion of study treatment
* Men must use a latex condom during sexual contact with fertile females during and for ≥ 28 days after completion of study treatment, even if a prior successful vasectomy was performed
* Stable neurological exam
* No serious medical condition or psychiatric illness that would preclude study participation
* No prior desquamating rash or allergic reaction ≥ grade 2 while taking thalidomide, lenalidomide, or structurally related compounds
* No peripheral neuropathy ≥ grade 2
* No active infection
* No uncontrolled hyper- or hypocalcemia, glycosemia, or thyroidism

PRIOR CONCURRENT THERAPY:

* No prior CC-4047
* More than 28 days since prior cytotoxic chemotherapy (42 days for nitrosoureas)
* At least 14 days since prior therapeutic radiotherapy
* More than 14 days since prior thalidomide, lenalidomide, or structurally related compounds
* More than 14 days since prior biological response modifier therapy
* Concurrent radiotherapy to treat pain associated with existing bone lesions during the extension phase of the study allowed provided < 10% of bone marrow is irradiated
* Concurrent systemic steroids for control of CNS primary tumor and/or metastases symptoms allowed provided dose is stable or decreasing AND patient is also taking low-dose aspirin and/or other platelet-active, anti-thrombotic medication during and for 30 days after completion of study treatment
* No other concurrent chemotherapy or immunotherapy
* No other concurrent investigational agents
* No concurrent hematopoietic growth factors during the treatment phase of the study
* No other concurrent anticancer agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2007-03; Primary Completion 2010-09 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | after initial 28 day cycle
  To determine the maximum tolerated dose (MTD) of daily CC-4047 in an initial 28-day cycle (21 days of CC-4047 followed by 7 days of no therapy) in subjects with advanced solid tumors (Cohort A).
Dose-limiting toxicity | Courses repeat every 28 days for up to 24 months in the absence of unacceptable toxicity.

SECONDARY OUTCOMES:
Tumor response as assessed by RECIST criteria | after every 2 courses (28 days/ course)
Duration of response | Courses repeat every 28 days for up to 24 months in the absence of disease progression.
Fetal hemoglobin levels as assessed thereafter | at baseline and every 28 days thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Matthew M. Cooney, MD, Study Chair — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center; Robert Dreicer, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio